CLINICAL TRIAL: NCT02121483
Title: An Open-label, Randomised, Multicentre, Single-dose, Parallel Group Trial to Evaluate Pharmacokinetics and Pharmacodynamics of Empagliflozin in Children and Adolescents From 10 to Less Than 18 Years of Age With Type 2 Diabetes Mellitus
Brief Title: Pharmacokinetic Single Dose Trial of Empagliflozin in Children and Adolescents With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.87; 2013-002304-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (3):
- empagliflozin high dose (Experimental): Patient to receive a high dose of empagliflozin
  Interventions: Drug: empagliflozin high dose
- empagliflozin medium dose (Experimental): Patient to receive a medium dose of empagliflozin
  Interventions: Drug: empagliflozin medium dose
- empagliflozin low dose (Experimental): Patient to receive a low dose of empagliflozin
  Interventions: Drug: empagliflozin low dose

INTERVENTIONS:
Drug: empagliflozin medium dose
  Arms: empagliflozin medium dose
Drug: empagliflozin high dose
  Arms: empagliflozin high dose
Drug: empagliflozin low dose
  Arms: empagliflozin low dose

SUMMARY:
The aim of the study is to generate pharmacokinetic and pharmacodynamic data to identify the safe-effective dose of empagliflozin in children and adolescents aged 10 to less than 18 years with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

* Children and adolescents with type 2 diabetes mellitus
* Insufficient glycaemic control (HbA1c <=10.5%) despite diet and exercise and/or metformin and/or stable basal or MDI insulin
* Negative for Islet Cell Antigen and Glutamic Acid Decarboxylase autoantibodies and fasting C-peptide levels >= 0.85 ng/ml
* BMI > 50th percentile for age and sex

Exclusion criteria:

* Uncontrolled hyperglycaemia with a glucose level > 240 mg/dl (> 13.3 mmol/l)
* History of acute metabolic decompensation such as diabetic ketoacidosis within 3 months before the screening visit with the exception of acute de-compensation at the time of type 2 diabetes diagnosis
* Treatment with weight reduction medications within 4 weeks before randomisation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (11):
- United States (5):
  - 1245.87.01013 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 1245.87.01004 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1245.87.01002 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1245.87.01012 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1245.87.01001 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
- 1245.87.33001 Boehringer Ingelheim Investigational Site, Lyon, France
- Israel (2):
  - 1245.87.97202 Boehringer Ingelheim Investigational Site, Beersheba
  - 1245.87.97203 Boehringer Ingelheim Investigational Site, Tel Litwinsky
- 1245.87.52001 Boehringer Ingelheim Investigational Site, Chihuahua City, Mexico
- South Africa (2):
  - 1245.87.27003 Boehringer Ingelheim Investigational Site, Bellville
  - 1245.87.27002 Boehringer Ingelheim Investigational Site, Pretoria

REFERENCES:
- [Derived] Bjornstad P, Laffel L, Tamborlane WV, Simons G, Hantel S, von Eynatten M, George J, Marquard J, Cherney DZI. Acute Effect of Empagliflozin on Fractional Excretion of Sodium and eGFR in Youth With Type 2 Diabetes. Diabetes Care. 2018 Aug;41(8):e129-e130. doi: 10.2337/dc18-0394. Epub 2018 Jun 25. No abstract available. PMID 29941496
- [Derived] Laffel LMB, Tamborlane WV, Yver A, Simons G, Wu J, Nock V, Hobson D, Hughan KS, Kaspers S, Marquard J. Pharmacokinetic and pharmacodynamic profile of the sodium-glucose co-transporter-2 inhibitor empagliflozin in young people with Type 2 diabetes: a randomized trial. Diabet Med. 2018 Aug;35(8):1096-1104. doi: 10.1111/dme.13629. Epub 2018 May 6. PMID 29655290

RESULTS

PARTICIPANT FLOW:
Groups:
- Empagliflozin 5mg: Single dose (1 tablet) of 5mg, empagliflozin, film-coated tablet administered orally.
- Empagliflozin 10mg: Single dose (1 tablet) of 10mg, empagliflozin, film-coated tablet administered orally.
- Empagliflozin 25mg: Single dose (1 tablet) of 25mg, empagliflozin, film-coated tablet administered orally.
Period: Overall Study
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Started | 9 | 8 | 10
Completed | 9 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all patients who were allocated trial medication and had received trial medication (empagliflozin).
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg | Total
Number analyzed (Participants) | 9 | 8 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.7 (2.0) | 14.5 (1.9) | 14.2 (2.1) | 14.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 7 | 18
  Male | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: AUC0-inf
Description: Area under the concentration-time curve of analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf).
Time Frame: Before drug administration (-0:30 hours (h)) and 0:30h, 1:00h, 1:30h, 2:00h, 4:00h, 8:00h, 12:00 (Day 1), 24:00 (Day 2), 34:00 (Day 2), 48:00 (Day 3) after drug administration.
Population: Pharmacokinetic Set (PKS): The PKS included all treated patients who provided at least 1 primary or secondary pharmacokinetic parameter for statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 9 | 8 | 10
nmol*h/L | 1150 (47.6) | 1430 (17.2) | 5060 (29.5)
Statistical Analysis 1: Comparison: Empagliflozin 5mg vs Empagliflozin 10mg vs Empagliflozin 25mg; Test type: Superiority or Other; Slope = 0.9490, 95% CI 2-sided [0.7276 to 1.1704], Standard Error of Mean 0.1075 — Dose proportionality was assessed based on a power model that describes the functional relationship between the dose and AUC0-inf. Based on the estimate for the slope parameter β, a 2-sided 95% confidence interval (CI) for the slope was computed

2. Primary Outcome: AUC0-tz
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 9 | 8 | 10
nmol*h/L | 1110 (49.9) | 1400 (17.1) | 4980 (29.1)
Statistical Analysis 1: Comparison: Empagliflozin 5mg vs Empagliflozin 10mg vs Empagliflozin 25mg; Test type: Superiority or Other; Slope = 0.9597, 95% CI 2-sided [0.7356 to 1.1838], Standard Error of Mean 0.1088 — Dose proportionality was assessed based on a power model that describes the functional relationship between the dose and AUC0-tz. Based on the estimate for the slope parameter β, a 2-sided 95% CI for the slope was computed

3. Primary Outcome: Cmax
Description: Maximum measured concentration in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 9 | 8 | 10
nmol/L | 159 (44.5) | 188 (50.2) | 602 (61.1)
Statistical Analysis 1: Comparison: Empagliflozin 5mg vs Empagliflozin 10mg vs Empagliflozin 25mg; Test type: Superiority or Other; Slope = 0.8554, 95% CI 2-sided [0.5504 to 1.1603], Standard Error of Mean 0.1481 — Dose proportionality was assessed based on a power model that describes the functional relationship between the dose and Cmax. Based on the estimate for the slope parameter β, a 2-sided 95% CI for the slope was computed

4. Primary Outcome: Tmax
Description: Maximum measured concentration in plasma (tmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 9 | 8 | 10
hours | 1.50 [0.95 to 7.92] | 1.25 [0.97 to 4.17] | 1.78 [0.50 to 4.00]

5. Primary Outcome: t1/2
Description: Terminal half-life in plasma (t1/2).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 9 | 8 | 10
hours | 6.92 (19.4) [5.46 to 8.90] | 7.35 (29.3) [4.51 to 10.90] | 7.80 (29.6) [4.93 to 11.10]

6. Secondary Outcome: Change From Baseline in Urinary Glucose Excretion (UGE) Over 24 h After Study Drug Intake
Description: Change from baseline in Urinary Glucose Excretion (UGE) over 24 h after study drug intake.
  For the changes from baseline in UGE on Day 1 (0 to 24 h postdose) , adjusted means per treatment group were to be calculated based on an ANCOVA including 'treatment' as a fixed effect and 'UGE at baseline' and 'FPG at baseline' as continuous covariates. Means presented are the adjusted means.
Time Frame: baseline and 24 hours
Population: Treated Set (TS) including patients with UGE data on both visits
Measure: Mean (Standard Error); unit: g/24h
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 8 | 8 | 10
g/24h | 53.1 (10.24) | 73.0 (10.14) | 87.4 (9.39)

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at 24 h After Study Drug Intake
Description: Change from baseline in Fasting Plasma Glucose (FPG) at 24h after study drug intake.
  For the change from baseline in FPG at 24 h postdose (in the morning of Day 2), adjusted means per treatment group were to be calculated based on an ANCOVA including 'treatment' as a fixed effect and 'FPG at baseline' as continuous covariate.
  Means presented are the adjusted means.
Time Frame: baseline and 24 hours
Population: Treated Set (TS) including patients with FPG data on both visits
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 7 | 8 | 10
mg/dL | -15.5 (6.53) | -16.6 (6.29) | -20.4 (5.68)

8. Secondary Outcome: Change From Baseline in 8-point Plasma Glucose Profile Over 24 h After Study Drug Intake
Description: Change from baseline in 8-point plasma glucose profile over 24h after study drug intake (as defined by change from baseline in Mean Daily Glucose (MDG) calculated at Day 1).
  For the changes from baseline in MDG on Day 1, adjusted means per treatment group were to be calculated based on an ANCOVA including 'treatment' as fixed effect and 'MDG at baseline' as continuous covariate.
  Means presented are the adjusted means.
Time Frame: baseline and 24 hours
Population: Treated Set (TS) including patients with plasma glucose profile data on both visits
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Number analyzed (Participants) | 5 | 4 | 7
mg/dL | -12.9 (7.95) | -6.5 (9.21) | -13.2 (7.00)

ADVERSE EVENTS:
Time Frame: All adverse events reported within 7 days following trial drug administration were considered on treatment, up to 8 days
Arm/Group | Empagliflozin 5mg | Empagliflozin 10mg | Empagliflozin 25mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 4/9 | 1/8 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 5mg (N=9) | Empagliflozin 10mg (N=8) | Empagliflozin 25mg (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.